CLINICAL TRIAL: NCT04361682
Title: Preoperative Systemic Inflammatory Biomarkers and Postoperative Day 1 Drain Amylase Value Predict Grade C Pancreatic Fistula After Pancreaticoduodenectomy: a Retrospective Single Center Experience
Brief Title: Preoperative Inflammatory Biomarkers and Postoperative Day 1 Drain Amylase Value Predict Pancreatic Fistula After Pancreaticoduodenectomy
Status: Completed | Type: Observational
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Damiano Caputo, Associate Professor of Surgery, Campus Bio-Medico University
Other Study IDs: 27/19 OSS ComEt CBM
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Pancreatic Fistula; Pancreas Cancer; Inflammatory Response
Keywords: Pancreatic Fistula; Pancreatic anastomoses; Surgical Drain Management; Inflammatory Biomarkers
MeSH Terms: conditions — Pancreatic Fistula; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgical Drain Management

SUMMARY:
Particularly, pancreatic fistula is the most common and serious complication after pancreaticoduodenectomy (PD) and is reported in up to 40% of cases. The aim of this retrospective single-center study was to investigate the utility of the combination of preoperative inflammation biomarkers (PIBs) with postoperative day 1 drains amylase (POD1-d.a.) levels in predicting grade C Pancreatic Fistula (PF).

DETAILED DESCRIPTION:
Data from a prospective collected database of 317 consecutive PDs performed at the University Campus Bio-Medico di Roma during the years 2005-2019, have been retrospectively analyzed. Local Ethical Committee approved the study.

Patients undergoing PD for periampullary neoplasms were included in the study. All patients underwent to PD with pancreaticojejunostomy reconstruction. Two surgical drains were always placed at the end of the surgery.

Data regarding PIBs, as full blood count including white blood cell (WBC) count, lymphocytes, neutrophils and platelets counts, neutrophil-to-lymphocyte ratio (NLR), derived neutrophil-to-lymphocyte ratio (d-NLR), platelet-to-lymphocyte ratio (PLR) and POD1-d.a. levels were collected and Positive Predictive Values (PPV) and Negative Predictive Values (NPV) were computed to investigate the probability to develop PF combining PIBs and drains amylase values.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent pancreaticoduodenectomy (PD) for periampullary neoplasms
* Patients underwent PD with pancreaticojejunostomy reconstruction.
* Patient with data of blood count in first postoperative day

Exclusion Criteria:

* None of the above criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According to the inclusion criteria, 227 patients were eligible for the study. The median age of all the series was 69 years (IQR= 60.25-74). Male patients were 131 (57.7%), the median BMI was 24.06 Kg/m2 (IQR= 22.15-27.59). Biochemical leak, grade B and grade C PF have been detected in 67/227 (29.5%), 21/227 (9.25%) and 22/227 (9.7%) of the cases, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Predictive value of PIBs and drains amylase values for Pancreatic Fistula (PF) | pre-intervention/ Day 1 after the intervention/up to discharge"
  Predictive Values (PPV) and Negative Predictive Values (NPV) were computed to investigate the probability to develop Pancreatic Fistula (PF) combining PIBs and Postoperative Day 1 Drain Amylase Value

IPD SHARING:
Plan to Share IPD: No